CLINICAL TRIAL: NCT00968344
Title: An Integrated Low-Volume Nutritional Countermeasure to Maintain Muscle Mass and Function During Space Exploration
Brief Title: Muscle Mass During Space Exploration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Space Biomedical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 09-121; MA02001 (Other Grant/Funding Number: NSBRI)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2017-12

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — Leucine; Alanine

STUDY DESIGN:
Intervention Model Description: Intervention: leucine
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leucine (Experimental): 3-4 g Leucine added to daily meals during bed rest
  Interventions: Dietary Supplement: Leucine
- Placebo (Placebo Comparator): 3-4 g Alanine added to daily meals during bed rest
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Leucine — 3-4g Leucine added to daily meals
  Arms: Leucine
Dietary Supplement: Alanine — Powered amino acid
  Arms: Placebo

SUMMARY:
The investigators will test the following hypotheses:

1. Bedrest will blunt the anabolic response to a mixed nutrient meal, facilitating a loss of muscle mass and functional capacity that is only partially restored during rehabilitation.
2. Enriching daily meals with leucine will promote protein synthesis and maintain the anabolic response to mixed nutrient meal ingestion. This will preserve lean muscle mass and function during bedrest and facilitate the recovery of functional and metabolic capacity during rehabilitation.

DETAILED DESCRIPTION:
Our long-term goal is to identify, prevent and remedy defects in the metabolic pathway that contribute to the loss of muscle mass and function during exposure to microgravity. Demographic data indicate that the average age of shuttle crew members has increased from 40.7 yrs in 1995 to 46.7 yrs in 2007 with an increasing number of astronauts over 50 yrs of age. We contend that the loss of muscle mass and function during spaceflight is facilitated by an age-associated, progressive impairment in the ability to mount an anabolic response to standard mixed nutrient meals. We propose that enriching daily meals with a low-volume leucine supplement will reduce the deleterious effects of microgravity on skeletal muscle and facilitate recovery during rehabilitation.

We will employ our established 14 day bed rest protocol to model the skeletal muscle unloading that occurs during microgravity. We will also examine recovery of muscle mass and functional capacity during a 7 day rehabilitation period. We will study 2 groups: CON (Bedrest/Recovery + Placebo; n=15), LEU (Bedrest/Recovery + Leucine; n=15). We will assess a) markers of translation initiation, b) muscle protein synthesis, c) muscle mass and body composition and d) strength and aerobic capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 45-60
2. Ability to sign informed consent

Exclusion Criteria:

1. Subjects with cardiac abnormalities considered exclusionary by the study physicians
2. Subjects with uncontrolled metabolic disease
3. A GFR <65 mL/min/1.73m2 or evidence of kidney disease or failure
4. Subjects with vascular disease or risk factors of peripheral atherosclerosis
5. Any history of hypo- or hyper-coagulation disorders. (e.g., Coumadin use or history of DVT or PE)
6. Subjects with chronically elevated systolic pressure >150 or a diastolic blood pressure > 100
7. Subjects with implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
8. Subjects with recently (6 months) treated cancer other than basal cell carcinoma
9. Any subject currently on a weight-loss diet or a body mass index > 30 kg/m2
10. Inability to abstain from smoking for duration of study
11. A history of > 20 pack per year smoking
12. Any subject that is HIV-seropositive or has active hepatitis
13. Recent anabolic or corticosteroids use (within 3 months)
14. Subjects with hemoglobin or hematocrit lower than accepted lab values
15. Agitation/aggression disorder
16. History of stroke with motor disability
17. A recent history (<12 months) of GI bleed
18. Any other condition or event considered exclusionary by the PI and faculty physician

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Paddon-Jones, PhD, Principal Investigator — The University of Texas Medical Branch at Galveston
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] English KL, Mettler JA, Ellison JB, Mamerow MM, Arentson-Lantz E, Pattarini JM, Ploutz-Snyder R, Sheffield-Moore M, Paddon-Jones D. Leucine partially protects muscle mass and function during bed rest in middle-aged adults. Am J Clin Nutr. 2016 Feb;103(2):465-73. doi: 10.3945/ajcn.115.112359. Epub 2015 Dec 30. PMID 26718415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2009-2014: we recruited and studied middle-aged men and women (45-60 years), representative of the ethnic makeup of the United States. Volunteers were recreationally active but athletically untrained.After providing written informed consent, volunteers were screened in the UTMB Institute for Translational Sciences-Clinical Research Center.
Groups:
- Leucine: 3-4 g Leucine added to daily meals during bed rest
  Leucine: crystalline amino acid
- Placebo: 3-4 g Alanine added to daily meals during bed rest
  Alanine: crystalline amino acid
Period: Overall Study
Arm/Group | Leucine | Placebo
Started | 20 (Includes screen fails) | 20 (Includes screen fails)
Completed | 10 | 9
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Population: Healthy community-dwelling men and women aged 45-60 y old participated in this randomized, double-blind, placebo controlled study. Volunteers were recreationally active but athletically untrained.
Groups:
- Total: Total of all reporting groups
Arm/Group | Leucine | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Screen fails not included
  Participants
    Female | 4 | 3 | 7
    Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Lean Leg Mass
Description: DEXA scan of both legs pre/post bed rest
Time Frame: At baseline prior to beginning bed rest and after 14 days of bed rest
Population: Healthy community-dwelling men and women aged 45-60 y
Measure: Mean (Standard Error); unit: g
Groups:
- Control Group: Subjects in the control group consumed a 3-4 g of alanine at each meal (an isonitrogenous control)
- Leucine (Intervention) Group: Subjects in the leucine group consumed 3-4 g of leucine at each meal during bed rest.
Arm/Group | Control Group | Leucine (Intervention) Group
Number analyzed (Participants) | 9 | 10
g | -1.2 (0.2) | -0.9 (0.1)

ADVERSE EVENTS:
Arm/Group | Leucine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No